CLINICAL TRIAL: NCT02461095
Title: Evaluation of a Treatment Algorithm for Patients With Patellofemoral Pain Syndrome: A Randomized Controlled Trial
Brief Title: Evaluation of a Treatment Algorithm for Patients With Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Mitchell Selhorst, Physical Therapist/Research Coordinator, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB15-00311
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Impairment based approach (Active Comparator): The intervention will address the patients impairments found during evaluation. Treatment will based on the Physical therapist evaluation and will be individualized to each patient.
  Interventions: Other: Impairment based approach
- PFPS algorithm (Experimental): The Patellofemoral Syndrome algorithm is designed to determine what deficits a patient may have and addressing these sequentially. This subgrouping first assesses a patient fear avoidance beliefs, flexibility, body mechanics, and then strength and functional ability. The reason for sequential treatment is that there is evidence that without adequate flexibility a patient will be unable to perform exercises with proper body mechanics, and without proper mechanics strengthening and functional activity can cause increased stress on the patellofemoral joint. Progression through each specific subgroup is based on objective goals. Once the patient has met these goals they are progressed to the next treatment subgroup until discharge.
  Interventions: Other: PFPS Algorithm approach

INTERVENTIONS:
Other: Impairment based approach — This intervention will consist of exercise, mechanics training, education, manual therapy and modalities. The treatment will address the impairments found during the evaluation. This approach is a typical individualized physical therapy treatment approach.
  Arms: Impairment based approach
Other: PFPS Algorithm approach — Physical Therapy treatment for Patellofemoral Pain Syndrome based upon a treatment algorithm that addresses patients: fear avoidance beliefs, flexibility, body mechanics, and strength. The exercises and treatments are individualized to each patient with the goals of low fear avoidance beliefs, flexibility, body mechanics, and strength and are performed in a sequential manner
  Arms: PFPS algorithm

SUMMARY:
Patients with PFPS demonstrate quadriceps and hip musculature weakness, altered lower extremity (LE) kinematics, and decreased LE flexibility. Psychosocial factors have also been identified as an important factor in patients with PFPS. The authors hypothesize that an ordered approach addressing each of these impairments sequentially will result in greater improvement in PFPS symptoms. The results of the investigators pilot study assessing the feasibility of using a sequential approach showed a full randomized controlled trial is warranted, the authors now plan to proceed with a full trial. The objective of this study is to assess the efficacy of a sequential approach in the treatment of Patellofemoral Pain Syndrome.

Methods: Patients will be randomized to a sequential treatment approach using a PFPS treatment algorithm (PFPS Algorithm) designed by the authors or typical physical therapy care. Due to the constant evaluation necessary no blinding will be performed. Patients will attend therapy two times per week for six weeks. Pain, Anterior Knee Pain Scale (AKPS), and Global Rating of Change (GROC) will be measured at evaluation and discharge, 3 month follow-up and 6 month follow-up.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) accounts for 25 to 40% of knee pain in young and active individuals. PFPS is described as anterior knee pain around the patella which is aggravated by activity, particularly activities that increase patellofemoral forces such as squatting, ascending or descending stairs, running, and jumping. It is common in adolescents and physically active adults. Females are more likely to experience PFPS than males. PFPS is a multi-factorial condition with no clear etiology and is considered a syndrome and not a diagnosis. Dye has described PFPS as one of the most difficult orthopedic conditions to manage.

Multiple theories exist regarding a cause for PFPS pain. A primary theory for the cause of PFPS is abnormal patellar tracking which results in excessive patellofemoral joint compressive forces. Many factors contributing to abnormal patellar tracking have been suggested including; hip and quadriceps weakness, delayed or diminished activation of vastus medialis obliquus, increased Q-angle, altered lower extremity mechanics and decreased lower extremity flexibility. Due to the number of suggested contributory factors to PFPS pain, a vast amount of interventions exist and are frequently used by clinicians. Although, physical therapy interventions have been shown to be effective over sham interventions, many individuals will have recurrent or chronic pain. Ninety-six percent of patients report having problems four years following their diagnosis of PFPS. A possible reason for the continued pain is that PFPS is a multi-factorial condition and the treatments may not address all of the contributing factors in each individual.

If all of the contributing factors for the patient's PFPS are identified, addressing all of these factors at once may not be the best approach. Performing hip strengthening prior to quadriceps strengthening results in decreased levels of pain with exercise. Individuals with reduced flexibility are more likely to have impaired lower extremity mechanics. Performing traditional lower extremity strengthening exercises when there is impaired lower extremity mechanics results in increased patellofemoral joint contact forces.

In an attempt to better treat individuals with PFPS, classification systems to subgroup patients with PFPS have been proposed, but their effectiveness has not been evaluated. An important clinical question with classification systems is what to do when a patient does not nicely fit into one subgroup. If a patient does not meet or meets the criteria for multiple subgroups, how is the patient treated? No evidence exists on the relative frequency with which patients with PFPS fall into each of these proposed subgroups and whether these subgroups are mutually exclusive.

The clinical classification systems reported in literature only address physical impairments. Psychosocial factors have also been identified as important when treating patients with PFPS. In a study by Piva et al. fear avoidance beliefs were the strongest predictor of outcomes for function and pain. Mental health status on the Medical Outcomes Short Form-36 is correlated with severity of patellofemoral symptoms in athletes. The results of these studies highlight the necessity of addressing psychosocial factors when treating PFPS.

Therefore, the authors have designed a new classification system (PFPS algorithm) for subgrouping patients based on the patient's clinical presentation. There are four subgroups in the new PFPS algorithm: Fear-Avoidance, Flexibility, Functional Malalignment, and Strengthening with function progression. The criteria and intervention of each subgroup is addressed sequentially over the episode of care. This classification system aims to address problems encountered if individuals meet the criteria for multiple subgroups. There is also a psychosocial component to address the needs of individuals with activity avoidance. The PFPS algorithm is goal-based, where meeting the criteria to pass through each subgroup is the focus of the treatment. Clinicians can provide whichever physical therapy intervention that allows an individual patient to meet the criteria of each subgroup. Interventions used in the PFPS algorithm are based on best available evidence, clinician's experience, and the patient's individual response to the intervention.

A pilot study assessing the feasibility of a full study assessing this algorithm and it effectiveness was performed previously by the study investigators (IRB13-00749). The primary aims of this pilot study were met. The therapists and clinic personnel successfully worked together to carry out all treatments required to conduct a future full scale randomized controlled trial. The ordered treatment approach used in the PFPS algorithm, addressing soft tissue tightness, altered lower extremity kinematics, neuromuscular deficits and psychosocial factors in a sequential manor, resulting in clinically significant improvements in Anterior Knee Pain Scale and Global Rating of Change scores. With minor changes to the protocol and outcome measures used, a full randomized controlled trial assessing the effectiveness of the PFPS algorithm was deemed feasible.

The primary objective of this study is to assess the efficacy of using a sequential treatment approach to treat patellofemoral pain syndrome.

Patient will be randomized into one of two treatment groups; either the PFPS algorithm or the control group which is an impairment based approach.

Impairment Based Approach:

The control group will be an impairment based approach with treatment focusing on impairments found during evaluation in the lower quarter. The evaluation of the lower quarter will assess motion, flexibility, strength and body mechanics. The joints of the lower quarter include the lumbar spine, hip, knee, ankle and foot. Specific attention will be paid to quadriceps and hip strength, hip and knee flexibility, and squatting, jumping, walking and running mechanics. Treatment will consist of 2 visits per week for 6 weeks. Treatments will last for 45-60 minutes. Exercises will be given for the patient to perform at home at the therapist discretion. Interventions will be individualized to the patient and will be at the therapist's discretion. Therapists can use treatments including but not limited to: exercise, manual therapy, taping and bracing, orthotics, modalities, and education. Home exercises will be given the therapist discretion consistent with standard care.

PFPS treatment algorithm:

The PFPS treatment algorithm is a objective goal driven treatment program. Treatment is at the therapist discretion with the objective to meet the requirements for each subgroup. Evidence from literature guides treatment to best meet these goals.

The first group within the classification system is Fear Avoidance, as research has shown that a change in fear-avoidance beliefs about physical activity is one of the best predictors for improved functional outcome.

The second group is Flexibility. This is the second group in the system because research shows that patients with decreased flexibility are unable to properly perform functional malalignment test. Also quadriceps length and gastrocnemius/soleus lengths are strongly associated with PFPS.

The third group is Functional Malalignment. This group assesses the patient's form with functional tasks. If the patient demonstrates impaired mechanics, time is spent with strengthening and motor control so that the patient will be able to strengthen and return to full function with proper technique.

The final group is Strengthening/Return to Function. This group will work strengthening of the lower quarter muscles with particular attention to the quadriceps, hip abductor and external rotators. This is also the time to progress the patient back to sport or functional activity.

-Fear Avoidance Belief Questionnaire (A score of 15 or greater on this questionnaire results in being give a PFPS fear avoidance booklet and treatment using a Cognitive Behavioral emphasis)

Primary Muscle Flexibility Requirements (Not meeting 1 of these flexibility measures results being placed into the flexibility subgroup)

* Quadriceps ≥ 130 degrees
* Gastrocnemius ≥ 12 degrees
* Soleus ≥ 20 degrees
* Weight Bearing Dorsiflexion ≥ 48 degrees

Secondary Muscle Flexibility (Having tightness in at least 3 of the following tests results in being placed into the flexibility subgroup)

* Thomas test
* Ober's Test
* Hamstring Straight Leg Raise ≥ 80 degrees
* Adductor Flexibility

Functional Malalignment (Score of great than 1 results in being placed into functional malalignment subgroup)

* Lateral Step Down test
* Single Leg Squat test

Strengthening/Functional Progression (A limb symmetry index score of >=90% for each of these test is used to determine adequate LE strength and function)

* Single Hop Test
* Triple Hop Test
* Crossover Hop for Distance test
* Timed Step Down test

ELIGIBILITY:
Inclusion Criteria:

-Clinical Diagnosis of Patellofemoral Pain Syndrome

Exclusion Criteria:

* Tenderness to palpation of patellar tendon, inferior pole of patella, or tibial tubercle as primary complaint
* Patient is pregnant or nursing
* Patient has other current lower extremity injuries
* History of patellar subluxation or dislocations
* History of knee surgery
* Inability to follow directions

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-06; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in Anterior Knee Pain Scale | Baseline, 3 weeks (18-24 days post-evaluation), 6 weeks (39-46 days post-evaluation), 3 months and 6 months
  Assessment of change of the Anterior Knee Pain Scale (AKPS). The AKPS is a self-reported 13 item questionnaire with discrete categories related to various levels of current knee function. Categories within each item are weighted, and responses are summed to provide an overall score of 0-100, with 100 representing no disability. The Anterior Knee Pain Scale is found to be valid and reliable in patients from 12-50 years of age presenting with anterior knee pain with a test-retest reliability of .95 (Watson, 2005). A change of 10 points represent the minimal clinical difference (Crossley, 2004).

SECONDARY OUTCOMES:
Change in Numeric Pain Rating Scale | Baseline, 3 weeks (18-24 days post-evaluation), 6 weeks (39-46 days post-evaluation), 3 months and 6 months
  The Numeric Pain rating scale asks the patient their highest pain in the last 24 hours. The Numeric Pain Rating Scale is a 0-10 scale subjectively assessing a patients perceived level of pain. With 0 on the scale = to no pain, and 10 = to the worst pain imaginable. The use of the Numerical Pain Rating Scale for assessing pain has been validated for use in PFPS patients and has been found to have a minimal detectable change of 1 points (Piva, 2009). The highest pain value is being used because of a floor effect was noted using average pain during the pilot study.
Global Rating of Change Scale (GROC) | Baseline, 3 weeks (18-24 days post-evaluation), 6 weeks (39-46 days post-evaluation), 3 months and 6 months
  The Global Rating of Change scale is a 15-point Likert type scale (-7 to +7). A score of 0 represents no change from initial injury, +7 represents a great deal better, and -7 represents a great deal worse. A score of +/- 3 represents a minimal clinical difference (Wang, 2011).

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Selhorst, DPT, Principal Investigator — Nationwide Childrens Hospital
Locations (4):
- United States (4):
  - Nationwide Children's Hospital Sports and Ortho PT East Broad, Columbus, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT Dublin, Dublin, Ohio
  - Nationwide Children's Hospital Sports and Ortho PT New Albany, New Albany, Ohio
  - Nationwide Children's Hospital Sports and Orthopedic PT Westerville location, Westerville, Ohio

REFERENCES:
- [Background] Powers CM, Bolgla LA, Callaghan MJ, Collins N, Sheehan FT. Patellofemoral pain: proximal, distal, and local factors, 2nd International Research Retreat. J Orthop Sports Phys Ther. 2012 Jun;42(6):A1-54. doi: 10.2519/jospt.2012.0301. Epub 2012 Jun 1. PMID 22660660
- [Background] Piva SR, Fitzgerald GK, Wisniewski S, Delitto A. Predictors of pain and function outcome after rehabilitation in patients with patellofemoral pain syndrome. J Rehabil Med. 2009 Jul;41(8):604-12. doi: 10.2340/16501977-0372. PMID 19565153
- [Background] Bolgla LA, Boling MC. An update for the conservative management of patellofemoral pain syndrome: a systematic review of the literature from 2000 to 2010. Int J Sports Phys Ther. 2011 Jun;6(2):112-25. PMID 21713229
- [Background] Wang YC, Hart DL, Stratford PW, Mioduski JE. Baseline dependency of minimal clinically important improvement. Phys Ther. 2011 May;91(5):675-88. doi: 10.2522/ptj.20100229. Epub 2011 Mar 3. PMID 21372203
- [Background] Piva SR, Gil AB, Moore CG, Fitzgerald GK. Responsiveness of the activities of daily living scale of the knee outcome survey and numeric pain rating scale in patients with patellofemoral pain. J Rehabil Med. 2009 Feb;41(3):129-35. doi: 10.2340/16501977-0295. PMID 19229444
- [Background] Watson CJ, Propps M, Ratner J, Zeigler DL, Horton P, Smith SS. Reliability and responsiveness of the lower extremity functional scale and the anterior knee pain scale in patients with anterior knee pain. J Orthop Sports Phys Ther. 2005 Mar;35(3):136-46. doi: 10.2519/jospt.2005.35.3.136. PMID 15839307
- [Background] Crossley KM, Bennell KL, Cowan SM, Green S. Analysis of outcome measures for persons with patellofemoral pain: which are reliable and valid? Arch Phys Med Rehabil. 2004 May;85(5):815-22. doi: 10.1016/s0003-9993(03)00613-0. PMID 15129407
- [Result] Selhorst M, Rice W, Degenhart T, Jackowski M, Tatman M. Evaluation of a treatment algorithm for patients with patellofemoral pain syndrome: a pilot study. Int J Sports Phys Ther. 2015 Apr;10(2):178-88. PMID 25883866